CLINICAL TRIAL: NCT04057495
Title: The Acute Effect of Mango Intake (Mangifera Indica L.) on Blood Pressure and Blood Glucose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Mango Board (Other); USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1453713
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Blood Pressure
Keywords: Blood glucose; Insulin
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- no mango intake (Placebo Comparator): No mango consumption on the study visit
  Interventions: Other: further fasting
- white bread with same amount of calorie as mango (Experimental): White bread consumption on the study visit
  Interventions: Other: white bread consumption
- mango consumption (Experimental): mango consumption on the study visit
  Interventions: Other: mango consumption

INTERVENTIONS:
Other: further fasting — 2 hours of fasting
  Arms: no mango intake
Other: white bread consumption — 113 grams of white bread consumption
  Arms: white bread with same amount of calorie as mango
Other: mango consumption — 330 grams of mango consumption
  Arms: mango consumption

SUMMARY:
In the current proposal the investigators seek to evaluate the acute effects of mango intake on blood pressure, blood glucose and insulin in postmenopausal women between 50 and 70 years old.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of mortality in the U.S, and aging is the largest risk factor for vascular diseases. Both male and female adults have increased risk for CVD as they age. For postmenopausal women, this risk is particularly elevated due to the loss of the protective effect of estrogen. It is evident that nutrition plays a crucial role in prevention of chronic diseases such as heart disease, stroke and cancer. Scientific evidence shows that high intake of plant-based food lowers the risk of CVD and many other chronic diseases.

Polyphenolic compounds in fruits and nuts have been the focus of extensive research regarding their potential to reduce risk for a number of chronic diseases. However, fruits and nuts vary largely in the type and amounts of phytonutrients they provide. Mango (Mangifera Idica L.), a commonly cultivated fruit worldwide, is rich in polyphenolic compounds such as gallic acid, mangiferin, quercetin glycosides, ferulic acid, and hydroxybenzoic acid. Many of those bioactive compounds have been found to have anti-diabetic and anti-inflammatory effects in cell models. For instance, mangiferin has been proved to effectively reducing glucose-induced endoplasmic reticulum stress by inhibiting IREα phosphorylation and ROS production in endothelial cells. However, it is unknown if the phytonutrients in mango will demonstrate a similar impact in humans. Therefore, the overall objective of this study is to investigate the effects of acute mango intake on blood pressure and blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female: 50-70 years
* Women: lack of menses for at least one year and FSH 23-116.3 mlU/mL
* Subject is willing and able to comply with the study protocols.
* Subject is willing participate in all study procedures
* BMI 25.0 - 40 kg/m2
* Weight ≥ 110 pounds

Exclusion Criteria:

* BMI ≥ 40 kg/m2
* Dislike or allergy for mango
* Self-reported use of daily anticoagulation agents including aspirin, NSAIDs
* Vegan, Vegetarians, food faddists or those consuming a non-traditional diet
* Alcohol consumption > 3 drinks/week (i.e. 1 bottle of beer, 1 glass of wine, and 1 shot of hard liquor)
* Fruit consumption ≥ 2 cups/day
* Vegetable consumption ≥ 3 cups/day for females
* Fatty Fish ≥ 3 times/week
* Coffee/tea ≥ 3 cups/day
* Dark chocolate ≥ 3 oz/day
* Self-reported restriction of physical activity due to a chronic health condition
* Self-reported chronic/routine high intensity exercise
* Self-reported diabetes
* Blood pressure ≥ 140/90 mm Hg
* Self-reported renal or liver disease
* Self-reported heart disease, which includes cardiovascular events and Stroke
* Abnormal Liver, CBC or Chemistry panels (laboratory values outside the reference range) if determined to be clinically significant by the study physician.
* Self-reported cancer within past 5 years
* Self-reported malabsorption

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | Baseline, 2 hours
  Changes in measures of blood pressure (mmHg) from baseline to two hours following fasting or consumption of white bread or mango.

SECONDARY OUTCOMES:
Change in blood glucose | Baseline, 2 hours
  Changes in blood glucose from baseline to two hours following fasting or consumption of white bread or mango.
Change in insulin levels | Baseline, 2 hours
  Changes in insulin from baseline to two hours following fasting or consumption of white bread or mango.

CONTACTS AND LOCATIONS:
Locations (1):
- Regal Human Nutrition Research Center, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No